CLINICAL TRIAL: NCT07119255
Title: The Effectiveness of Pharmacopuncture With Platelet-Rich Plasma (PRP) as a Treatment for Chronic Neck Pain in Cervical Myofascial Syndrome Related to the Upper Trapezius Muscle
Brief Title: Effectiveness of PRP Pharmacopuncture for Chronic Neck Pain in Cervical Myofascial Syndrome of the Upper Trapezius
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Irma Nareswari, MD, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-05-0695
Record Dates: First submitted 2025-07-28; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Neck Pain; Myofascial Pain Syndrome
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Pharmacopuncture (Experimental): Participants in the PRP pharmacopuncture arm will receive a single administration of platelet-rich plasma (PRP) via intramuscular injection at acupuncture points corresponding to chronic neck pain in cervical myofascial syndrome in the upper trapezius muscle.
  Interventions: Procedure: PRP Pharmacopuncture
- Placebo Pharmacopuncture (Placebo Comparator): Participants in the placebo pharmacopuncture arm will receive a single administration of normal saline via intramuscular injection at acupuncture points corresponding to chronic neck pain in cervical myofascial syndrome in the upper trapezius muscle.
  Interventions: Procedure: Placebo Pharmacopuncture

INTERVENTIONS:
Procedure: PRP Pharmacopuncture — Participants in the PRP pharmacopuncture arm will receive a single administration of platelet-rich plasma (PRP) via intramuscular injection at acupuncture points corresponding to chronic neck pain in cervical myofascial syndrome in the upper trapezius muscle.
  Arms: PRP Pharmacopuncture
Procedure: Placebo Pharmacopuncture — Participants in the placebo pharmacopuncture arm will receive a single administration of normal saline via intramuscular injection at acupuncture points corresponding to chronic neck pain in cervical myofascial syndrome in the upper trapezius muscle.
  Arms: Placebo Pharmacopuncture

SUMMARY:
The goal of this clinical trial is to learn whether pharmacopuncture with Platelet-Rich Plasma (PRP) is effective for treating chronic neck pain in cervical myofascial syndrome related to the upper trapezius muscle. The main questions it aims to answer are:

1. Is pharmacopuncture with Platelet-Rich Plasma (PRP) effective in reducing chronic neck pain in patients with cervical myofascial syndrome related to the upper trapezius muscle?
2. Does PRP pharmacopuncture improve functional outcomes and quality of life in these patients?
3. Are there any adverse effects associated with PRP pharmacopuncture in this context?

Researchers will compare PRP pharmacopuncture to normal saline pharmacopuncture (placebo) to evaluate whether PRP provides greater effectiveness in reducing chronic neck pain in cervical myofascial syndrome related to the upper trapezius muscle.

Participants will:

* Receive a single session of pharmacopuncture therapy
* Undergo evaluations at week 2, week 4, and week 8 after the intervention

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate the effectiveness of PRP pharmacopuncture in patients with chronic neck pain in cervical myofascial syndrome related to the upper trapezius muscle. Participants are 60 males/females aged 18-59 years. They will be divided into two groups: (1) PRP pharmacopuncture and (2) Normal saline (placebo) pharmacopuncture. Each participant will receive a single pharmacopuncture treatment. Therapy efficacy will be assessed at week 2, week 4, and week 8 after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 59 years.
* Experiencing neck pain for more than 3 months (chronic).
* Neck pain classified as Grade I to III according to the Neck Pain Task Force classification.
* Presence of referred pain pattern on physical examination consistent with the distribution of the upper trapezius muscle.
* Visual Analogue Scale (VAS) score between 30 and 70 mm (out of 100 mm) during activity (e.g., daily activities or light exercise).
* Willing to participate in the study until completion and has signed the informed consent form.

Exclusion Criteria:

* Hemoglobin level <13 g/dL for males or <12 g/dL for females.
* Platelet count <150,000/μL.
* Presence of fever (≥37.5°C).
* Diagnosis of fibromyalgia.
* Structural abnormalities of the cervical spine other than degenerative changes, such as fractures, cervical spine injuries, space-occupying lesions (SOL), infections, neoplasms, or systemic diseases confirmed by radiographic imaging.
* History of cervical spine surgery.
* Presence of tumors, wounds, or skin infections at the needle insertion site.
* Diagnosed with blood disorders or currently taking anticoagulant or antiplatelet medications.
* History of hypersensitivity reactions to acupuncture (e.g., metal allergy, severe atopy, keloids, or other skin hypersensitivities).
* Uncontrolled cardiovascular disease or diabetes mellitus.
* History of pharmacopuncture therapy to the upper trapezius muscle within the past 6 months.
* Use of anti-inflammatory medication within the past 2 weeks.
* Currently pregnant or breastfeeding.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Biomarker parameters | before treatment (baseline) and 4 weeks after treatment
  The serum concentration of interleukin-1 beta (IL-1β) and vascular endothelial growth factor (VEGF) will be measured as outcome biomarkers to evaluate inflammatory and angiogenic responses following the intervention.

SECONDARY OUTCOMES:
Visual Analogue Scale | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  Pain intensity will be assessed using a 100 mm horizontal visual analogue scale, where 0 mm indicates "no pain" and 100 mm indicates "worst imaginable pain." Participants will mark the point on the line that best represents their perceived pain intensity.
Pressure Pain Threshold | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  Using the minimum force applied which induces pain, measured with algometer
Neck Disability Index | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  A questionnaire for measuring self-rated disability due to neck pain
Perceived Stress Scale | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  psychological instrument for measuring the perception of stress. It assesses the degree to which individuals perceive situations in their lives as stressful over the past month. The scale consists of 10 items, each rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("very often"). Total scores range from 0 to 40, with higher scores indicating greater perceived stress.
Pain Catastrophizing Scale | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  a validated self-report questionnaire designed to assess catastrophic thinking related to pain. It consists of 13 items divided into three subscales: rumination, magnification, and helplessness. Each item is rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("all the time"), with total scores ranging from 0 to 52. Higher scores reflect greater levels of pain catastrophizing.
Short-Form 12 Health Survey | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  designed to assess health-related quality of life (HRQoL) across two main domains: physical and mental health.
Cervical Range of Motion | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  To evaluate the degree of movement in cervical flexion, extension, lateral flexion, and rotation using a goniometer or inclinometer.
Craniovertebral Angle | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  To assess head and neck posture, measured from lateral photographic analysis.
Size of Myofascial Trigger Point Nodules | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  The diameter (in millimeters) of hypoechoic nodules identified at active trigger point sites will be measured using B-mode ultrasound. Measurements will be taken in both longitudinal and transverse planes.
Resistive Index | before treatment (baseline), 2 weeks, 4 weeks, and 8 weeks after treatment
  The resistive index of the local blood flow surrounding the trigger point area will be assessed using color Doppler and spectral Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - RSCM

IPD SHARING:
Plan to Share IPD: No